Statistical plan for Historically Controlled Trial of Corticosteroids in Young Boys With Duchenne Muscular Dystrophy

Statistics will be performed with Excel (Microsoft Inc.) and GraphPad Prism (GraphPad Software, La Jolla, CA). P-values will all 2-tailed. A p value of <0.05 will interpreted as showing statistical significance. Mann Whitney U will be used for non-parametric data.

Analysis of data will be performed in two ways. First, the change over one year in the Treated Cohort will be compared to the previously published Historical Control Cohort (HCC). Second, repeated measures (paired t- tests) were used to analyze each boy's performance over his own baseline.